CLINICAL TRIAL: NCT00409994
Title: A Clinical Trial Testing Rapamycin, an mTOR-inhibitor, in Combination With Preoperative Radiotherapy in Operable Rectum Cancer: a Phase I and Phase II Study
Brief Title: Safety Study of Rapamycin Administered Before and During Radiotherapy to Treat Rectum Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-16
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Rectum Cancer
Keywords: Colorectal cancer; M-tor inhibitor; Rapamycin
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rapamycine (Experimental): rapamycine 6 mg dd
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — dosis escalation: 2/4/6 mg rapamycin tablets, once daily during 13 days
  Other Names: Sirolimus

SUMMARY:
Investigating the safety and the activity of Rapamycin, administered before and during preoperative radiotherapy in patients with an operable colorectal carcinoma. The phase I dose escalation study will be performed in three steps (2, 4 and 6 mg). Patients entered in phase II will follow the same tolerable treatment regimen as patients in phase I study.

DETAILED DESCRIPTION:
Treatment regimen Phase I A daily dose of Rapamycin will be taken during 13 days. At step 1 a dose of 2 mg will be given once a day; at step 2 a dose of 4 mg will be given once a day; at step 3 a dose of 6 mg will be given once a day.

Preoperative radiotherapy (5x 5 Gy) will be administered at day 8-12, followed by TME-surgery at day 15.

Phase II A daily dose of 6 mg Rapamycin will be taken for 14 days (unless the optimal dose found in the phase I study is lower).

Preoperative radiotherapy (5x 5 Gy) will be administered at day 9-15, followed by TME-surgery 7-8 weeks post RT.

Sample size Phase I dose-escalation study Minimum 3 eligible patients per step, maximum 6 eligible patients per step. Phase II A total of 47 patients will be entered in this part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven rectum cancer
* UICC TNM I-III
* WHO performance status 0-2
* Less than 10% weight loss the last 6 months
* No recent (< 3 months) severe cardiac disease
* Normal serum bilirubin and serum creatinin

Exclusion Criteria:

* Concurrent chemotherapy with radiation
* History of prior pelvis radiotherapy
* Recent (<3 months) myocardial infarction
* Uncontrolled infectious disease
* Concurrent medication known as inhibitors of CYP3A4 susceptible to increase Rapamycin blood concentrations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-09; Primary Completion 2018-08-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Phase I: Incidence of severe postoperative complications (grade IV or grade V), | within the first 6 weeks after surgery
assessed according to CTCv3.0 | within the first 6 weeks after surgery
Phase II: Tumour blood flow assessed CT-PET + CTp | day 64

SECONDARY OUTCOMES:
Phase I:Incidence of other acute toxicity, assessed according to CTCv 3.0 | within the first 6 weeks after surgery
Activation status of mTor related and dependent molecules in the tumour | within the first 6 weeks after surgery
Phase II:Maximum standardised Uptake Value (SUV) of 18F-FDG, assessed bij PET-CT-scan | day 64
Phase II:Incidence of acute side effects of rapamycin, assessed according to CTCv 4.0 | day 8, 15, 22, 36, 50 and 64

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Buijsen, MD PhD, Principal Investigator — Maastricht Radiation Oncology
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Limburg, Netherlands